CLINICAL TRIAL: NCT06323239
Title: Stereotactic Body Radiotherapy (SBRT) and Low-dose Radiotherapy (LDRT) Combined With Programmed Death 1 (PD-1) Antibody and Chemotherapy in Recurrent/Metastatic Nasopharyngeal Carcinoma: A Prospective, Single-arm, Phase II Clinical Trial
Brief Title: SBRT and LDRT Combined With PD-1 Antibody and Chemotherapy in r/m Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Dr. Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT/LDRT+PD-1+GP for r/mNPC
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: SBRT; Low-dose radiotherapy; PD-1 antibody; Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy; toripalimab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+LDRT+PD-1+Chemotherapy (Experimental): Patients will receive SBRT and LDRT one day before the GP chemotherapy and PD-1 antibody (six cycles), then followed by PD-1 antibody until progressive disease, intolerable toxicity, withdrawal of consent or a maximum of 2 year treatment.
  Interventions: Radiation: SBRT; Radiation: Low-dose Radiotherapy (LDRT); Drug: Toripalimab; Drug: Gemcitabine; Drug: Cisplatin; Radiation: IMRT

INTERVENTIONS:
Radiation: SBRT — SBRT for metastatic lesions
Radiation: Low-dose Radiotherapy (LDRT) — LDRT for metastatic lesions
Drug: Toripalimab — 6 cycles for combined therapy. Toripalimab maintenance for 1 year.
Drug: Gemcitabine — 6 cycles for combined therapy.
Drug: Cisplatin — 6 cycles for combined therapy.
Radiation: IMRT — IMRT for primary lesion

SUMMARY:
This is a prospective, single-arm, phase II clinical trial. The purpose of this study is to evaluate the efficacy and adverse effect of SBRT and LDRT combined with programmed death 1 (PD-1) antibody and chemotherapy in recurrent/metastatic nasopharyngeal carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as recurrence/metastatic NPC
* Histopathological diagnosis of NPC(WHO II/III)
* ECOG 0-1 point
* No treatment to r/mNPC, such as radiotherapy, chemotherapy, immunotherapy or biotherapy;
* No contraindications to immunotherapy and chemoradiotherapy;
* At least one lesion could receive SBRT safely;
* Subject must have a measurable target lesion based on RECIST v1.1;
* Adequate marrow function: WBC count ≥ 3×10E9/L, NE count ≥ 1.5×10E9/ L, HGB ≥ 90g/L, PLT count ≥ 100×10E9/L;
* Adequate liver function: ALT/AST ≤ 2.5×ULN, TBIL ≤ 2.0×ULN;
* Adequate renal function: BUN/CRE ≤ 1.5×ULN or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
* Take effective contraceptions during and three months after treatment;
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* Allergic to monoclonal antibodies, any PD-1 antibody components, gemcitabine and cisplatin;
* Unexplained fever > 38.5 #, except for tumor fever;
* Have active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy);
* Have a known history of human immunodeficiency virus (HIV), active Hepatitis B (HBV-DNA ≥10E3copiers/ml) or hepatitis C virus (HCV) antibody positive;
* Have New York Heart Association (NYHA) class 3 or 4, unstable angina, myocardial -infarction within 1 year, or clinically meaningful arrhythmia that requires treatment; Have known allergy to large molecule protein products or any compound of study therapy;
* Pregnant or breastfeeding;
* Prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical cancer, and papillary thyroid carcinoma;
* Have received a live vaccine within 30 days of planned start of study therapy Has psychiatric drug or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
* Any other condition, including mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 12 months
  Defined as the time from randomization to the first occurrence of disease progression as determined according to RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival | up to 12 months
  Defined as the time from randomization to death from any cause.
Objective Response Rate | up to 12 months
  The percentage of patients with CR and PR assessed according to RECIST v1.1.
Disease Control Rate | up to 12 months
  The proportion of patients who have achieved complete response, partial response and stable disease according to RECIST v1.1.
Adverse Events | up to 12 months
  All adverse event or serious adverse event that occurred during the study period according to CTCAE v 4.03
QoL | up to 12 months
  Assessed by EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, MD. PhD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China